CLINICAL TRIAL: NCT00405665
Title: Pilot Study of the Short Term Safety and Efficacy of Inhaled L-arginine in Patients With Cystic Fibrosis
Brief Title: The Short Term Safety and Efficacy of Inhaled L-arginine in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000009282
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; L-Arginine; Pediatrics; pulmonary function
MeSH Terms: conditions — Cystic Fibrosis | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: L-arginine
- 2 (Experimental)
  Interventions: Drug: L-arginine

INTERVENTIONS:
Drug: L-arginine — Group 1 will receive the active treatment followed by the inactive treatment. The active treatment phase will consist of L-arginine 250 mg/ml dispensed in 2.2 ml vials, from which the patient will take 2ml (500mg) and dilute with 3ml of sterile water to give 5ml of a 100mg/ml solution. Dosing in the inactive treatment phase will consist of a placebo of similar osmolarity and appearance will be formulated and dosed in a similar fashion. It will consist of 2.2ml vials of 1110mmol/L hypertonic saline. Again, the patient will take 2ml and dilute with 3ml of sterile water to give a 445mmol/L solution which has similar tonicity (10%) to the L-arginine. Both treatment phases will be administered by inhalation with a PARI eFLOW device.
  Arms: 1
Drug: L-arginine — Group 2 will receive the inactive treatment followed by the active treatment.
  Arms: 2

SUMMARY:
The objective of this trial is to determine the safety and effect on pulmonary function of 14 days of inhaled L-arginine versus placebo administered over a period of 14 days in a cohort of CF patients.

DETAILED DESCRIPTION:
Despite the inflammatory nature of lung disease in CF, nitric oxide (NO) formation as well as the expression of NOS2 has been found to be decreased in CF airways. While the reasons for impaired airway NO formation remain incompletely understood, there is evidence that low NO formation contributes to lung pathophysiology in CF. Constitutive endogenous formation of Nitric oxide (NO) in airways is thought to play a role in neurotransmission, smooth muscle relaxation and bronchodilation. Previous animal experiments have shown that the addition of L-arginine, the precursor of enzymatic NO formation, resulted in a significantly greater relaxation of tracheas. There is also evidence that a single dose of inhaled L-arginine improves pulmonary function in CF. In this study we will assess the effect of L-arginine inhalation on lung function, nitric oxide formation, airway inflammation and bacterial infection in CF patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as defined by two or more clinical features of CF and a documented sweat chloride concentration > 60 mEq/L and/or two well characterized disease causing CFTR gene mutations
* 14 years of age and older at enrollment
* Clinically stable at enrollment
* Ability to comply with medication use, study visits and study procedures
* FEV1 % predicted > 40% < 80 % as calculated by reference equations

Exclusion Criteria:

* Respiratory culture positive for: B. cepacia complex within past year or at screening
* Use of systemic corticosteroids within 30 days of screening
* Use of intravenous antibiotics or oral quinolones within 14 days of screening
* History of biliary cirrhosis, portal hypertension, or splenomegaly
* Other major organ dysfunction
* History of lung transplantation or currently on lung transplant list
* Supplemental oxygen therapy
* Oxygen saturation < 95 % on room air
* Positive pregnancy test at screening
* Investigational drug use within 30 days of screening
* History of alcohol, illicit drug or medication abuse within 1 year of screening
* Acute respiratory symptoms
* Inability to take any form of bronchodilator
* Wheezing at the time of study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 (in liters) from baseline | At the end of the 14 day treatment period
Adverse events such as gastrointestinal complaints, wheezing, hepatitis or shortness of breath | 70 weeks

SECONDARY OUTCOMES:
Change in FVC and change in FEV25-75 from baseline to completion of the 2 week treatment period. | Will be measured at the end of the 14 day treatment period
Change in exhaled nitric oxide (FeNO) | 70 days
Changes in inflammatory markers in sputum from baseline including neutrophils (sputum), neutrophil elastase (sputum) and interleukin (IL)-8 concentrations (sputum). | Will me measured at the end of the 14 day treatment period
Changes in sputum concentrations of L-arginine metabolites | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Wark P, McDonald VM, Smith S. Nebulised hypertonic saline for cystic fibrosis. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD001506. doi: 10.1002/14651858.CD001506.pub5. PMID 37319354
- [Derived] Grasemann H, Tullis E, Ratjen F. A randomized controlled trial of inhaled L-arginine in patients with cystic fibrosis. J Cyst Fibros. 2013 Sep;12(5):468-74. doi: 10.1016/j.jcf.2012.12.008. Epub 2013 Jan 14. PMID 23333044